CLINICAL TRIAL: NCT04440930
Title: Can White Tea Prevent Oral Mucositis in Patients Receiving Neoadjuvant or Adjuvant Treatment With Paclitaxel for Breast Cancer? A Randomized Trial
Brief Title: White Tea for Prevention of Chemotherapy Induced Mucositis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vejle Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: WHITE TEA
Record Dates: First submitted 2020-06-18; First posted 2020-06-22 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-09

CONDITIONS: Oral Mucositis
Keywords: mucositis; mouth; paclitaxel
MeSH Terms: conditions — Stomatitis; Mucositis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- White tea (Experimental)
  Interventions: Other: White tea
- Salt water with soda (Active Comparator)
  Interventions: Other: Salt water with soda

INTERVENTIONS:
Other: White tea — Mouthwash with white tea five to six times a day for nine weeks
  Arms: White tea
Other: Salt water with soda — Mouthwash with salt water and soda eight to ten times a day for nine weeks
  Arms: Salt water with soda

SUMMARY:
The aim of this study is to determine the effectiveness of mouthwash with white tea in the prevention of paclitaxel induced oral mucositis in women with breast cancer.

DETAILED DESCRIPTION:
Oral mucositis is a common side effect from paclitaxel treatment. It can be very painful and compromise nutrition and oral hygiene, and it may increase the risk of infection. Although oral mucositis is a common side effect to chemotherapy, no available treatment is yet available that can effectively prevent or treat oral mucositis.

Based on the knowledge that white tea has anti-inflammatory, anti-oxidant and anti-microbial effect, the current study aims to assess the effect of mouth wash with white tea on paclitaxel induced oral mucositis in women with breast cancer.

This study is a phase II randomized controlled trial in which eligible patients will be allocated to a control group (CG) and a study group (SG). The CG will use salt water with soda for mouthwash eight to ten times a day and the SG will use white tea for mouthwash five to six times a day.

ELIGIBILITY:
Inclusion Criteria:

* Woman with breast cancer
* Planned neoadjuvant or adjuvant paclitaxel treatment
* Age ≥ 18 years
* Understand and speak Danish
* Written and orally informed consent

Exclusion Criteria:

- Palliative treatment with paclitaxel

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2020-09-02 (Actual); Primary Completion 2023-03-28 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Incidence of oral mucositis grade 2 or higher as measured by the Revised Oral Assessment Guide. | up to nine weeks
  Nine categories are included in the Revised Oral Assessment Guide tool: voice, lips, mucous, tongue, gums, teeth, saliva, denture and swallowing. Each category is described and rated according to a score of 1 (healthy) to 3 (severe problems).

SECONDARY OUTCOMES:
Frequency of daily mouthwashes | once a week over a period of nine weeks
  Number of daily mouthwashes will be registered
Frequency of daily tooth brushings | once a week over a period of nine weeks
  Number of daily tooth brushings will be registered
Pain intensity in the oral cavity as measured on the Numeric Rating Scale (NRS). | Once a week over a period of nine weeks
  Numeric Rating Scale 0-10; 0=no pain, 10=worst possible pain
Date of onset of oral mucositis grade 2 or higher as measured by Revised Oral Assessment Guide. | Once a week until oral mucositis occurs up to nine weeks
  Nine categories are included in the Revised Oral Assessment Guide tool: voice, lips, mucous, tongue, gums, teeth, saliva, denture and swallowing. Each category is described and rated according to a score of 1 (healthy) to 3 (severe problems).

CONTACTS AND LOCATIONS:
Overall Officials: Erik H Jakobsen, MD, Study Chair — Vejle Hospital
Locations (1):
- Department of Oncology, Vejle Hospital, Vejle, Denmark